CLINICAL TRIAL: NCT01327495
Title: Dose Response Effects of Exogenous Testosterone on the Prostate and Comparison With Effects on Body Composition (Short Title: PROS-2)
Brief Title: PROS-2 Dose Response Effects of Exogenous Testosterone on the Prostate
Acronym: PROS-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephanie T. Page, Professor Department of Medicine, Division of Metabolism, Endocrinology and Nutrition, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39738; 1R01AG037603-01 (NIH)
Record Dates: First submitted 2011-03-21; First posted 2011-04-01 (Estimated); Results first posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Androgen replacement in men
MeSH Terms: interventions — Testosterone; Gels; acyline; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1: Placebo (Placebo Comparator): Placebo acyline every 2 weeks for two weeks + daily placebo gel x 12 weeks
  Interventions: Other: placebo acyline; Other: placebo gel
- Arm 2:1.25g Testosterone (Active Comparator): Acyline (300µg/kg every two weeks) + testosterone 1% gel 1.25 g daily x 12 weeks
  Interventions: Drug: Testosterone 1% gel 1.25 g; Drug: Acyline
- Arm 3: 2.5g Testosterone (Active Comparator): Acyline (300µg/kg every two weeks) + testosterone 1% gel 2.5 g daily x 12 weeks
  Interventions: Drug: Testosterone 1% gel 2.5 g; Drug: Acyline
- Arm 4: 5g Testosterone (Active Comparator): Acyline (300µg/kg every two weeks) + testosterone 1% gel 5.0 g daily x 12 weeks
  Interventions: Drug: Testosterone 1% gel 5.0 g; Drug: Acyline
- Arm 5: 10g Testosterone (Active Comparator): Acyline (300µg/kg every two weeks) + testosterone 1% gel 10 g daily x 12 weeks
  Interventions: Drug: testosterone 1% gel 10 g; Drug: Acyline
- Arm 6: 15g Testosterone (Active Comparator): Acyline (300µg/kg every two weeks) + testosterone 1% gel 15 g daily x 12 weeks
  Interventions: Drug: testosterone 1% gel 15 g; Drug: Acyline

INTERVENTIONS:
Other: placebo acyline — Placebo acyline subcutaneous injection every 2 weeks
  Other Names: placebo
  Arms: Arm 1: Placebo
Other: placebo gel — daily placebo testosterone gel applied transdermally x 12 weeks
  Other Names: placebo
  Arms: Arm 1: Placebo
Drug: Testosterone 1% gel 1.25 g — testosterone 1% gel 1.25 g daily applied transdermally x 12 weeks
  Other Names: Androgel
  Arms: Arm 2:1.25g Testosterone
Drug: Testosterone 1% gel 2.5 g — Testosterone 1% gel 2.5 g daily applied transdermally x 12 weeks
  Other Names: Androgel
  Arms: Arm 3: 2.5g Testosterone
Drug: Testosterone 1% gel 5.0 g — Testosterone 1% gel 5.0 g daily applied transdermally x 12 weeks
  Other Names: Androgel
  Arms: Arm 4: 5g Testosterone
Drug: testosterone 1% gel 10 g — Testosterone 1% gel 10 g daily applied transdermally x 12 weeks
  Other Names: Androgel
  Arms: Arm 5: 10g Testosterone
Drug: testosterone 1% gel 15 g — Testosterone 1% gel 15 g daily applied transdermally x 12 weeks
  Other Names: Androgel
  Arms: Arm 6: 15g Testosterone
Drug: Acyline — 300 ug/kg subcutaneous injection every 2 weeks
  Other Names: GNRH antagonist
  Arms: Arm 2:1.25g Testosterone; Arm 3: 2.5g Testosterone; Arm 4: 5g Testosterone; Arm 5: 10g Testosterone; Arm 6: 15g Testosterone

SUMMARY:
The investigators will conduct a three-month, randomized, placebo-controlled trial comparing the effects of increasing doses of androgen supplementation with Testosterone (T) gel on the prostate in healthy men who are treated with acyline to block gonadal androgen production.

DETAILED DESCRIPTION:
The investigators overall goals are (i) to determine the relationship between serum and prostate tissue hormone concentrations in men in response to increasing doses of exogenous androgens; (ii) to determine the impact that alterations in serum and tissue testosterone concentrations have on prostate epithelial cell function and phenotype; and (iii) to determine the relationships between prostatic androgens and alterations in the tissue microenvironment. The investigators will perform a study in healthy, middle-aged men to address the following Specific Aims:

Specific Aims: To compare the dose-response relationships between serum testosterone and intraprostatic androgens and androgen action, and serum testosterone and anabolic activity in healthy, middle-aged men.

Hypothesis: The investigators hypothesize that very low levels of serum testosterone will lower concentrations of intraprostatic testosterone and dihydrotestosterone (DHT). However, when serum testosterone concentrations are within or even above the normal range there will be no significant increases in intraprostatic testosterone and dihydrotestosterone. In contrast, the investigators expect that anabolic activity will increase with increasing concentrations of circulating testosterone.

Secondarily, the investigators hypothesize that increasing levels of serum testosterone beyond the low normal range will have little impact on androgen action within the prostate.

Approach: The investigators will conduct a randomized, placebo-controlled trial in healthy men who are medically castrated and administered one of five different doses of testosterone gel (Androgel) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

In good health, without severe systemic illness (i.e., renal, liver, cardiac or lung disease, cancer, insulin dependent diabetes)

* Male between the ages of 25 and 55 years old
* Able to understand and comply with protocol instructions and requirements
* International Prostate Symptom Score (IPSS) <11
* Agrees to not donate blood during the study
* Normal serum total T, LH, FSH, urine analysis, COMP, CBC and sperm count

Exclusion Criteria:

* History of, or current breast cancer or prostate cancer
* Clinically significant findings on digital rectal exam such as nodules, areas of induration or any other malignancy or abnormal prostate ultrasound
* History of invasive therapy for BPH
* Current or past treatment with a 5α-reductase inhibitor
* History of drug or alcohol abuse within the past 12 months
* History of a bleeding disorder or anticoagulation
* Skin disease that might interfere with T-gel absorption
* Participation in another drug study in the past 3 months
* A first-degree relative (i.e. father, brother) with a history of prostate cancer
* History of infertility or desire for fertility within 6 months, or current pregnant female partner
* Weight >320 pounds or BMI > 40
* PSA Level > 2.1

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Page, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thirumalai A, Cooper LA, Rubinow KB, Amory JK, Lin DW, Wright JL, Marck BT, Matsumoto AM, Page ST. Stable Intraprostatic Dihydrotestosterone in Healthy Medically Castrate Men Treated With Exogenous Testosterone. J Clin Endocrinol Metab. 2016 Jul;101(7):2937-44. doi: 10.1210/jc.2016-1483. Epub 2016 May 12. PMID 27172434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy males, 25-55 years old, were recruited via advertisement: flyers and newspaper ads at the University of Washington.
Pre-assignment Details: 98 screened. 28 screen fails (or did not finish screen). 8 subjects dropped out prior to drug start. 62 subjects started drug. 7 subjects dropped after drug start/pre-drug finish. 2 dropped after finishing study drug, but prior to prostate biopsy. 2 subjects dropped from analysis for non-compliance. 51 completed entire study, included in analysis.
Groups:
- Arm 1 (Placebo Acyline & Placebo T Gel ): Placebo acyline every 2 weeks for two weeks + daily placebo gel x 12 weeks
  placebo acyline: Placebo acyline subcutaneous injection every 2 weeks
  placebo gel: daily placebo testosterone gel applied transdermally x 12 weeks
- Arm 2 (Acyline & 1.25g Testosterone Gel): Acyline (300µg/kg every two weeks) + testosterone 1% gel 1.25 g daily x 12 weeks
  Testosterone 1% gel 1.25 g: testosterone 1% gel 1.25 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 3 (Acyline & 2.5g Testosterone Gel): Acyline (300µg/kg every two weeks) + testosterone 1% gel 2.5 g daily x 12 weeks
  Testosterone 1% gel 2.5 g: Testosterone 1% gel 2.5 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 4 (Acyline & 5g Testosterone Gel): Acyline (300µg/kg every two weeks) + testosterone 1% gel 5.0 g daily x 12 weeks
  Testosterone 1% gel 5.0 g: Testosterone 1% gel 5.0 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 5 (Acyline & 10g Testosterone Gel): Acyline (300µg/kg every two weeks) + testosterone 1% gel 10 g daily x 12 weeks
  testosterone 1% gel 10 g: Testosterone 1% gel 10 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 6 (Acyline & 15g Testosterone Gel): Acyline (300µg/kg every two weeks) + testosterone 1% gel 15 g daily x 12 weeks
  testosterone 1% gel 15 g: Testosterone 1% gel 15 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
Period: Overall Study
Arm/Group | Arm 1 (Placebo Acyline & Placebo T Gel ) | Arm 2 (Acyline & 1.25g Testosterone Gel) | Arm 3 (Acyline & 2.5g Testosterone Gel) | Arm 4 (Acyline & 5g Testosterone Gel) | Arm 5 (Acyline & 10g Testosterone Gel) | Arm 6 (Acyline & 15g Testosterone Gel)
Started | 10 | 11 | 10 | 9 | 11 | 11
Completed | 8 (1 dropped due to decreased libido & energy, 1 dropped due to too much pain with acyline injections) | 9 (1 subject declined prostate biopsy & no-showed to final visit, 1 subject dropped d/t elevated LFTs.) | 8 (1 withdrawn due to injection AE. 1 drop-out (declined prostate biopsy and final visit).) | 9 | 8 (1 dropped out pre drug finish, 2 non-compliant subjects dropped) | 9 (1 subject withdrawn d/t elevated LFTs, 1 dropped out d/t ski accident)
Not Completed | 2 | 2 | 2 | 0 | 3 | 2
Not completed — Adverse Event | 2 | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 62 subjects started treatment, 11 dropped after drug start & pre-study exit visit (7 dropped post-drug start but pre-drug finish, 2 dropped after drug finish but pre-prostate biopsy, 2 dropped for non-compliance). 51 participants included in the analysis.
Groups:
- Arm 1: Placebo acyline every 2 weeks for two weeks + daily placebo gel x 12 weeks
  placebo acyline: Placebo acyline subcutaneous injection every 2 weeks
  placebo gel: daily placebo testosterone gel applied transdermally x 12 weeks
- Arm 2: Acyline (300µg/kg every two weeks) + testosterone 1% gel 1.25 g daily x 12 weeks
  Testosterone 1% gel 1.25 g: testosterone 1% gel 1.25 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 3: Acyline (300µg/kg every two weeks) + testosterone 1% gel 2.5 g daily x 12 weeks
  Testosterone 1% gel 2.5 g: Testosterone 1% gel 2.5 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 4: Acyline (300µg/kg every two weeks) + testosterone 1% gel 5.0 g daily x 12 weeks
  Testosterone 1% gel 5.0 g: Testosterone 1% gel 5.0 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 5: Acyline (300µg/kg every two weeks) + testosterone 1% gel 10 g daily x 12 weeks
  testosterone 1% gel 10 g: Testosterone 1% gel 10 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Arm 6: Acyline (300µg/kg every two weeks) + testosterone 1% gel 15 g daily x 12 weeks
  testosterone 1% gel 15 g: Testosterone 1% gel 15 g daily applied transdermally x 12 weeks
  Acyline: 300 ug/kg subcutaneous injection every 2 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Total
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9 | 51
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 45 [34 to 48] | 45 [41 to 46] | 46 [39 to 51] | 34 [30 to 44] | 42 [33 to 47] | 51 [50 to 54] | 44 [35 to 50]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 8 | 9 | 8 | 9 | 8 | 9 | 51
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg^m2] | 28 [26 to 33] | 28 [25 to 33] | 26 [24 to 28] | 25 [25 to 27] | 25 [22 to 28] | 26 [25 to 28] | 26 [25 to 29]
Testosterone Level [Median (Inter-Quartile Range); unit: ng/dL] | 450 [315 to 516] | 448 [345 to 509] | 554 [462 to 730] | 419 [387 to 505] | 482 [429 to 591] | 452 [396 to 536] | 459 [390 to 530]
DHT Level [Median (Inter-Quartile Range); unit: ng/dL] | 36 [27 to 47] | 37 [24 to 44] | 43 [39 to 59] | 39 [18 to 49] | 49 [44 to 55] | 36 [28 to 53] | 40 [28 to 52]
Lutenizing Hormone [Median (Inter-Quartile Range); unit: mIU/mL] | 3.5 [3 to 4.5] | 5 [4 to 6] | 4 [2 to 5.5] | 3 [3 to 4] | 4 [4 to 5] | 3 [3 to 5] | 4 [3 to 5]
FSH [Median (Inter-Quartile Range); unit: mIU/mL] | 5.5 [4 to 8.5] | 4 [3 to 6] | 5 [3 to 6] | 5 [3 to 6] | 5.5 [5 to 7] | 7 [4 to 8] | 5 [4 to 7]
Hematocrit [Median (Inter-Quartile Range); unit: %] | 43 [42 to 45] | 43 [41 to 44] | 43 [42 to 44] | 44 [41 to 46] | 45 [42 to 45] | 43 [41 to 44] | 43 [41 to 45]
Prostate Specific Antigen (PSA) [Median (Inter-Quartile Range); unit: ng/dL] | 0.80 [0.61 to 0.91] | 0.71 [0.66 to 0.88] | 1.09 [0.75 to 1.25] | 0.74 [0.34 to 0.86] | 0.67 [0.41 to 0.91] | 0.69 [0.35 to 0.91] | 0.75 [0.42 to 0.96]
Prostate volume [Median (Inter-Quartile Range); unit: cm^3] | 20 [16 to 22] | 19 [13 to 23] | 17 [17 to 21] | 17 [14 to 18] | 17 [14 to 20] | 19 [15 to 19] | 18 [14 to 21]
International Prostate Symptom Score (IPSS) [Median (Inter-Quartile Range); unit: units on a scale] — 0-7 mildly symptomatic, 8-19 moderately symptomatic, 20-35 severely symptomatic
  units on a scale | 2.5 [1.5 to 3] | 1 [1 to 3] | 2 [0 to 4.25] | 0 [0 to 1] | 1.5 [0 to 3] | 2 [1 to 3] | 2 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Prostate Tissue DHT Concentrations After Treatment
Description: To measure intraprostatic dihydrotestosterone [DHT] levels
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Groups:
- Arm 1/Placebo Acyline Inject & Placebo Testosterone Gel: Placebo acyline subcutaneous injection every 2 weeks for 12 weeks & daily placebo testosterone (T) gel applied transdermally for 12 weeks.
- Arm 2 Acyline Inject Every 2 Weeks & Daily T 1% Gel 1.25g: Acyline (300ug/kg) subcutaneous injection every 2 weeks for 12 weeks & daily 1% testosterone (T) gel 1.25g applied transdermally for 12 weeks.
- Arm 3 Acyline Inject Every 2 Weeks & Daily T 1% Gel 2.5: Acyline (300ug/kg) subcutaneous injection every 2 weeks for 12 weeks & daily 1% testosterone (T) gel 2.5g applied transdermally for 12 weeks.
- Acyline Inject Every 2 Weeks & Daily T 1% Gel 5g: Acyline (300ug/kg) subcutaneous injection every 2 weeks for 12 weeks & daily 1% testosterone (T) gel 5g applied transdermally for 12 weeks.
- Acyline Inject Every 2 Weeks & Daily T 1% Gel 10g: Acyline (300ug/kg) subcutaneous injection every 2 weeks for 12 weeks & daily 1% testosterone (T) gel 10g applied transdermally for 12 weeks.
- Acyline Inject Every 2 Weeks & Daily T 1% Gel 15g: Acyline (300ug/kg) subcutaneous injection every 2 weeks for 12 weeks & daily 1% testosterone (T) gel 15g applied transdermally for 12 weeks.
Arm/Group | Arm 1/Placebo Acyline Inject & Placebo Testosterone Gel | Arm 2 Acyline Inject Every 2 Weeks & Daily T 1% Gel 1.25g | Arm 3 Acyline Inject Every 2 Weeks & Daily T 1% Gel 2.5 | Acyline Inject Every 2 Weeks & Daily T 1% Gel 5g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 10g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 15g
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 4.05 [3.75 to 4.62] | 4.26 [2.7 to 5.57] | 2.99 [2.57 to 3.79] | 3.88 [3.61 to 4.476] | 4.12 [2.04 to 6.30] | 5.11 [4.4 to 8.69]

2. Primary Outcome: Serum Testosterone
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm 1/Placebo Acyline Inject & Placebo Testosterone Gel | Arm 2 Acyline Inject Every 2 Weeks & Daily T 1% Gel 1.25g | Arm 3 Acyline Inject Every 2 Weeks & Daily T 1% Gel 2.5 | Acyline Inject Every 2 Weeks & Daily T 1% Gel 5g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 10g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 15g
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/mL | 4.6 [3.1 to 5.0] | 1.9 [1.3 to 3.8] | 3.4 [2.5 to 4.4] | 3.5 [2.9 to 6.4] | 6.1 [2.7 to 9.9] | 7.7 [5.3 to 10.9]

3. Primary Outcome: Dihydrotestosterone (DHT)
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm 1/Placebo Acyline Inject & Placebo Testosterone Gel | Arm 2 Acyline Inject Every 2 Weeks & Daily T 1% Gel 1.25g | Arm 3 Acyline Inject Every 2 Weeks & Daily T 1% Gel 2.5 | Acyline Inject Every 2 Weeks & Daily T 1% Gel 5g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 10g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 15g
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/mL | 0.3 [0.3 to 0.5] | 0.6 [0.3 to 0.7] | 0.9 [0.5 to 1.2] | 1.0 [0.7 to 1.2] | 1.5 [0.6 to 2.5] | 1.8 [1.0 to 3.6]

4. Primary Outcome: Prostate Tissue Testosterone Concentrations After Treatment
Description: To measure intraprostatic testosterone levels
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1/Placebo Acyline Inject & Placebo Testosterone Gel | Arm 2 Acyline Inject Every 2 Weeks & Daily T 1% Gel 1.25g | Arm 3 Acyline Inject Every 2 Weeks & Daily T 1% Gel 2.5 | Acyline Inject Every 2 Weeks & Daily T 1% Gel 5g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 10g | Acyline Inject Every 2 Weeks & Daily T 1% Gel 15g
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 0.3 [0.2275 to 0.535] | 0.13 [0.11 to 0.24] | 0.125 [0.1075 to 0.165] | 0.18 [0.15 to 0.35] | 0.195 [0.1275 to 0.77] | 0.3 [0.22 to 1.72]

5. Secondary Outcome: Prostate Specific Antigen
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/dL | 0.82 [0.57 to 0.97] | 0.48 [0.44 to 0.62] | 0.61 [0.39 to 0.81] | 0.58 [0.41 to 0.78] | 0.52 [0.43 to 0.67] | 0.76 [0.50 to 1.2]

6. Secondary Outcome: Prostate Volume
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: cm^3
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
cm^3 | 19 [18 to 22] | 18 [14 to 22] | 19 [15 to 21] | 15 [14 to 17] | 16 [15 to 20] | 20 [16 to 20]

7. Secondary Outcome: International Prostate Symptom Score (IPSS)
Description: IPSS score: 0-7 mildly symptomatic, 8-19 moderately symptomatic, 20-35 severely symptomatic
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
units on a scale | 1 [0 to 2] | 2 [1 to 3] | 2.5 [1.5 to 5.25] | 0 [0 to 0] | 2.5 [1.5 to 7.75] | 4 [1 to 10]

8. Other Pre Specified Outcome: 17-OHPreg
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 1.19 [1.06 to 1.44] | 1.25 [0.93 to 2.07] | 1.23 [0.92 to 2.04] | 1.05 [1.01 to 1.89] | 1.02 [0.94 to 1.45] | 1.36 [1.29 to 1.47]

9. Other Pre Specified Outcome: 17-OHP
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 0.05 [0.04 to 0.06] | 0.05 [0.05 to 0.06] | 0.05 [0.04 to 0.05] | 0.05 [0.04 to 0.05] | 0.05 [0.04 to 0.05] | 0.05 [0.04 to 0.07]

10. Other Pre Specified Outcome: Androstenedione
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 0.16 [0.10 to 0.33] | 0.11 [0.10 to 0.18] | 0.12 [0.09 to 0.15] | 0.13 [0.12 to 0.15] | 0.18 [0.15 to 0.28] | 0.14 [0.12 to 0.22]

11. Other Pre Specified Outcome: Androsterone
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 0.17 [0.14 to 0.21] | 0.15 [0.12 to 0.22] | 0.12 [0.08 to 0.14] | 0.17 [0.11 to 0.24] | 0.17 [0.12 to 0.43] | 0.21 [0.17 to 0.23]

12. Other Pre Specified Outcome: DHEA
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 29.3 [19.1 to 42.0] | 26.2 [13.5 to 35.8] | 22.1 [16.2 to 30.1] | 26.8 [26.0 to 29.2] | 24.4 [23.0 to 28.2] | 18.6 [14.7 to 22.0]

13. Other Pre Specified Outcome: Pregnenolone
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 28.7 [23.6 to 33.8] | 29.5 [21.3 to 36.4] | 32.7 [23.3 to 51.2] | 32.4 [28.6 to 45.5] | 27.9 [17.4 to 37.6] | 23.9 [18.1 to 25.0]

14. Other Pre Specified Outcome: Progesterone
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 8 | 9
ng/g | 0.09 [0.06 to 0.20] | 0.08 [0.06 to 0.09] | 0.06 [0.04 to 0.09] | 0.08 [0.07 to 0.13] | 0.09 [0.08 to 0.12] | 0.07 [0.07 to 0.08]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from day 1 through the end of study, Week 18. After the screening period, 12 weeks of treatment commenced for subjects who met inclusion/exclusion criteria, followed by a 6 week recovery period.
Description: The 62 subjects who started study drugs on Day 0 were monitored for adverse events. Nine subjects were discontinued prior to study end. Two subjects were not included in data analysis due to medication non-compliance. Hence, while there were 51 subjects included in the analysis, 62 subjects (all who started study drugs) were monitored for adverse events.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/9 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 7/10 | 8/11 | 6/10 | 7/9 | 10/11 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=11) | Arm 3 (N=10) | Arm 4 (N=9) | Arm 5 (N=11) | Arm 6 (N=11)
Abnormal liver funtion tests (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction to Acyline (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort at injection site (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes/night sweats (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood changes (irritability) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased libido (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased libido (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased energy, fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Semen changes (decreased ejaculation volume (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin changes (acne, rash at site of T gel (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Nipple discomfort (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexually transmitted disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea, vomiting, abnormal bowl movements (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory infection/symptoms (Infections and infestations) | 2 (2) | 2 (5) | 0 (0) | 5 (5) | 2 (2) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Injuries/accidents (General disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Blood in semen (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruise at injection site (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes